CLINICAL TRIAL: NCT01568814
Title: Efficacy and Tolerability of Morning (AM) Only Low Volume (2L) PEG With Low Residue Test Meals Versus High Volume (4L) Split-dose (PM/AM) PEG Bowel Preparation With Standard Meals: A Prospective Randomized, Investigator Blinded Trial
Brief Title: Low Volume PEG With Low Residue Test Meals Versus High Volume Split-dose PEG Bowel Preparation
Acronym: LOWPEG
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Inje University (Other)
Responsible Party: Principal Investigator, Eun Hee Seo, MD, Principal investigator, Inje University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 1.0-A2012
Record Dates: First submitted 2012-03-29; First posted 2012-04-02 (Estimated); Last update posted 2012-04-03 (Estimated); Status verified 2012-01

CONDITIONS: Bowel Preparation; Colonoscopy
Keywords: colonoscopy; bowel preparation; polyethylene glycol; low residue meal

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- High volume PEG (Placebo Comparator): Patients who are scheduled colonoscopy ingest high volume PEG(4L) for bowel preparation.
  Interventions: Drug: high volume PEG
- Low volume PEG with low residual meals (Active Comparator): Patients who are scheduled colonoscopy ingest low volume PEG(2L) and have a prepackaged low residual meals for bowel preparation.
  Interventions: Drug: Low volume PEG

INTERVENTIONS:
Drug: Low volume PEG — low volume polyethylene glycol 2 liter one time
  Arms: Low volume PEG with low residual meals
Drug: high volume PEG — high volume polyethylene glycol 4 lilter split-dosing 2L/2L two times
  Arms: High volume PEG

SUMMARY:
Morning only low volume PEG with low reside meals may enhance patient tolerability and have similar bowel cleansing efficacy compared to standard method using high volume split-dose PEG with standard diet.

DETAILED DESCRIPTION:
We aimed to evaluate the efficacy and tolerability of bowel preparation protocols with low volume PEG and low residue meals PEG compared to conventional high volume (4L) split-dose and standard diet.

Entry criteria: Entry criteria: Adult outpatients and inpatients (18-85 years of age) who undergo colonoscopy for screening, cancer surveillance or with gastrointestinal symptoms, other symptoms

Primary Outcome: Quality of bowel preparation (Ottawa scale) Secondary Outcome: Tolerability (preparation completion, side effect), acceptance, willingness

ELIGIBILITY:
Inclusion Criteria:

* Adult outpatients and inpatients (18-85 years of age) who undergo colonoscopy for screening, cancer surveillance or with gastrointestinal symptoms, other symptoms

Exclusion Criteria:

* Age under 18 years
* Pregnancy
* Breast feeding
* Prior history of surgical large bowel resection
* Severe medical condition such as severe cardiac
* Hepatic, renal failure (creatinine ≥ 3.0mg/dL (normal 0.8-1.4))
* Drug addiction or major psychiatric illness
* Suspected bowel obstruction or ileus
* Allergy to PEG
* Refusal of consent to participate in the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2012-01; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Quality of bowel preparation | 2 months
  Quality of bowel preparation is assessed using Ottawa bowel preparation scale.

SECONDARY OUTCOMES:
Tolerability | 2 months
  Tolerability of bowel preparation regimen is assessed by patient questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Haeundae Paik Hospital, Inje University School of Medicine, Busan, South Korea